CLINICAL TRIAL: NCT01951729
Title: The Effects of GIP and/or Xenin-25, With and Without Atropine, on Insulin Secretion in Humans With Pre-diabetes
Brief Title: The Role of Cholinergic Signaling for Mediating the Effects of GIP and/or Xenin-25 on Insulin Secretion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 08-0861E
Record Dates: First submitted 2013-09-18; First posted 2013-09-27 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Pre-diabetes
Keywords: Blood sugar; GIP; Xenin-25; Cholinergic Signaling; Atropine; Insulin; Glucagon; Pancreatic polypeptide
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — Atropine; xenin 25; Albumins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pre-diabetes (Experimental): Otherwise healthy individuals exhibiting hemoglobin A1c levels between 6.0% - 7.0%
  Interventions: Drug: Control; Drug: Xenin-25 without atropine; Drug: GIP without atropine; Drug: Placebo with atropine; Drug: Xenin-25 with atropine; Drug: GIP with atropine; Drug: GIP plus Xenin-25 without atropine; Drug: GIP plus Xenin-25 with atropine

INTERVENTIONS:
Drug: Control — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes. The study is finished at 240 minutes.
  Starting at 0 minutes, an intravenous infusion of saline containing 1% human albumin will continue for 240 minutes.
  Other Names: No Peptide or Atropine
Drug: Xenin-25 without atropine — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes. The study is finished at 240 minutes.
  Following a priming dose from 0-10 minutes, xenin-25 (in saline containing 1% human albumin) will be administered at a constant dose of 4 pmoles/kg/min until 240 minutes.
  Other Names: xenin without atropine
Drug: GIP without atropine — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes. The study is finished at 240 minutes.
  Following a priming dose from 0-10 minutes, GIP (in saline containing 1% human albumin) will be administered at a dose of 4 pmoles/kg/min until 240 minutes.
Drug: Placebo with atropine — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes. The study is finished at 240 minutes.
  Following a priming dose from -30 to -28 minutes, atropine will be administered at a constant dose of 0.3 mg/m2/hour until 240 minutes.
  Other Names: Albumin (no peptide) with atropine
Drug: Xenin-25 with atropine — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes. The study is finished at 240 minutes.
  Following a priming dose from 0-10 minutes, xenin-25 (in saline containing 1% human albumin) will be administered at a dose of 4 pmoles/kg/min until 240 minutes.
  Following a priming dose from -30 to -28 minutes, atropine will be administered at a constant dose of 0.3 mg/m2/hour until 240 minutes.
  Other Names: xenin and atropine
Drug: GIP with atropine — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes. The study is finished at 240 minutes.
  Following a priming dose from 0-10 minutes, GIP (iin saline containing 1% human albumin) will be administered at a dose of 4 pmoles/kg/min until 240 minutes.
  Following a priming dose from -30 to -28 minutes, atropine will be administered at a constant dose of 0.3 mg/m2/hour until 240 minutes.
  Other Names: GIP and atropine
Drug: GIP plus Xenin-25 without atropine — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes. The study is finished at 240 minutes.
  Following a priming dose from 0-10 minutes, GIP and xenin-25 will each be administered at a dose of 4 pmoles/kg/min until 240 minutes.
  Other Names: GIP plus xenin without atropine
Drug: GIP plus Xenin-25 with atropine — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes. The study is finished at 240 minutes.
  Following a priming dose from 0-10 minutes, GIP and xenin-25 will each be administered at a dose of 4 pmoles/kg/min until 240 minutes.
  Following a priming dose from -30 to -28 minutes, atropine will be administered at a constant dose of 0.3 mg/m2/hour until 240 minutes.
  Other Names: GIP plus xenin with atropine

SUMMARY:
Glucose-dependent insulinotropic polypeptide (GIP) is a hormone produced in the intestine. It is released immediately after meal ingestion and increases insulin release. This, in turn, helps reduce blood glucose levels. This circuit does not work properly in humans with type 2 diabetes mellitus (T2DM).

We have previously shown that a peptide called xenin-25 can amplify the effects of GIP on insulin secretion in humans. However, xenin-25 no longer does this when humans develop T2DM. Thus, it is important to understand how xenin-25 works in humans without T2DM so we know why it does not work in humans with T2DM.

Acetylcholine is molecule produced by specific types of nerves. The effects of acetylcholine can be blocked by a drug called atropine. We have previously shown in mice that atropine prevents the ability of xenin-25 to increase the effects of GIP on insulin release. The purpose of this clinical trial is to determine if atropine also blocks the effects of xenin-25 in humans without T2DM. If it does, then impaired acetylcholine signaling may be one of the reasons humans develop T2DM and it could be possible to develop drugs that bypass this defect and increase insulin release in humans with T2DM.

DETAILED DESCRIPTION:
Glucose-dependent insulinotropic polypeptide (GIP) is a hormone produced in the intestine. It is released immediately after meal ingestion and increases insulin release. This, in turn, helps reduce blood glucose levels. This circuit does not work properly in humans with type 2 diabetes mellitus (T2DM).

We have previously shown that a peptide called xenin-25 can amplify the effects of GIP on insulin secretion in humans. However, xenin-25 no longer does this when humans develop T2DM. Thus, it is important to understand how xenin-25 works in humans without T2DM so we know why it does not work in humans with T2DM.

Acetylcholine is molecule produced by specific types of nerves. The effects of acetylcholine can be blocked by a drug called atropine. We have previously shown in mice that atropine prevents the ability of xenin-25 to increase the effects of GIP on insulin release. The purpose of this clinical trial is to determine if atropine also blocks the effects of xenin-25 in humans without T2DM. If it does, then impaired acetylcholine signaling may be one of the reasons humans develop T2DM and it may be possible to develop drugs that bypass this defect and increase insulin release in humans with T2DM.

To conduct this study, we will enroll humans with pre-diabetes since they respond very well to xenin-25. Potential subjects will first be checked to see if they do have pre-diabetes and also to verify that they can safely participate in the study. Once enrolled, subjects will come for 8 different visits, each separated by about 3 weeks. On each visit, the subject will be given an intravenous infusion of glucose such that blood glucose levels slowly increase over a 4 hour period. On separate occasions, the participant will also receive an infusion GIP alone, xenin-25 alone, GIP plus xenin-25, or placebo. Each of these 4 infusions will be conducted with and without an infusion of atropine (thus- the 8 visits). Blood glucose and insulin levels, as well as a host of other hormones, will be measured during each of the study visits. A comparison of the results will tell us if the effects of xenin-25 on insulin release are mediated by acetylcholine in humans.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be able to consent for their own participation (no mental impairment affecting cognition or willingness to follow study instructions).
* Otherwise healthy volunteers that have borderline diabetes or impaired glucose tolerance.
* Women of childbearing potential must be currently taking/using an acceptable method of birth control. A pregnancy test will be done at the beginning of each visit. Any woman with a positive pregnancy test will be removed from the study.
* Willingness to complete all required visits.

Exclusion Criteria:

* Lacks cognitive ability to sign the consent or follow the study directions.
* Women unwilling to use an acceptable method of contraception during the course of the study, or who are currently breast-feeding.
* Volunteers with a history of Acute Pancreatitis.
* Volunteers with a history of cancer (except for skin cancer).
* Volunteer with a history of Chronic Pancreatitis and/or risk factors for chronic pancreatitis including hypertriglyceridemia, hypercalcemia and/or the presence of gallstones.
* Volunteers with a history of gastrointestinal disorders, particularly related to gastric motility/emptying such as gastric bypass
* Subjects taking medications known to affect glucose tolerance.
* Anemia
* Significant systemic illness including heart, kidney, inflammatory, liver, or malignant disease requiring medications.
* Narrow-angle glaucoma
* Obstructive uropathy including benign prostatic hypertrophy, pyloric stenosis, myasthenia gravis
* Asthma
* hyperthyroidism
* angina and cardiac arrhythmias including heart block
* Subjects unwilling to allow the use of human albumin in the preparation of the peptides.
* Unwillingness to allow blood glucose level adjustment (if needed) with IV insulin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Insulin secretion rates during each treatment. | 3 years

SECONDARY OUTCOMES:
Plasma glucose levels during each treatment. | 3 years
Plasma glucagon levels during each treatment. | 3 years
Plasma pancreatic polypeptide levels during each treatment. | 3 years

OTHER OUTCOMES:
Plasma GIP levels during each treatment | 3 years
Plasma xenin-25 levels during each treatment. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Burton M Wice, PhD, Principal Investigator — Washington University School of Medicine; Dominic Reeds, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States